CLINICAL TRIAL: NCT06027086
Title: A Phase 1b/2 Study of Glutamine Antagonist DRP-104 in Combination With Durvalumab in Patients With Advanced Stage Fibrolamellar Hepatocellular Carcinoma (FLC)
Brief Title: DRP-104 (Glutamine Antagonist) in Combination With Durvalumab in Patients With Advanced Stage Fibrolamellar Carcinoma (FLC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Dracen Pharmaceuticals, Inc. (Industry); Fibrolamellar Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J23107; IRB00388561 (Other: Johns Hopkins Medical Institution)
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Fibrolamellar Hepatocellular Carcinoma
Keywords: Fibrolamellar Carcinoma (FLC); Durvalumab; DRP-104 (glutamine antagonist); Immunotherapy; Anti PD-L1; PD-L1; Carcinoma; Glutamine antagonist
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma; Carcinoma | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab and DRP-104 (Experimental)
  Interventions: Drug: Durvalumab; Drug: DRP-104

INTERVENTIONS:
Drug: Durvalumab — Patients will receive treatment on Day 1 of each cycle. Durvalumab (1500 mg) will be administered IV on Day 1 of each cycle every 28 days.
  Other Names: IMFINZI
Drug: DRP-104 — Patients will receive treatment twice a week of each cycle. DRP-104 (145 mg,125mg, 105mg, 85mg or 65mg) will be administered subcutaneous injection twice a week of each 28 day cycle.
  After the first cycle of treatment the study drug may be shipped to the patient's home for future cycles of administration if patients or caregiver can demonstrate at least two observed independent injections of DRP-104 prior to home administration.

SUMMARY:
The purpose of this study is to determine whether the combination of subcutaneous DRP-104 in combination with intravenous Durvalumab is safe and yields a clinically compelling antitumor activity measured as based on objective response rate (ORR, assessed by RECIST 1.1). Secondary objectives include progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed FLC (Fibrolamellar Carcinoma) that is metastatic or unresectable.
* Presence of DNAJB1-PRKACA fusion transcript, assessed by RNA-sequencing, DNA-sequencing, or in situ hybridization in the archival tissue.
* Must have demonstrated radiographic progression on prior or current immunotherapy.
* Age ≥ 12 years.
* Patients < 18 years old must have a body weight ≥ 40 kg.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
* Patients must have adequate kidney and liver function defined by study-specified laboratory tests.
* Must have measurable disease per RECIST 1.1
* Willingness to provide tissue and blood samples for mandatory translational research.
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test.
* For both Women and Men, must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Must have had chemotherapy or other systemic therapy or radiotherapy, as follows:

  * Patients who have had chemotherapy, biological cancer therapy, or radiation 21 days prior to the first dose of study drug.
  * Patients who have had surgery within 28 days of dosing of investigational agent, excluding minor procedures.
  * Patients who have received other approved or investigational agents or device within 21 days of the first dose of study drug.
* Patients who have not recovered from acute adverse events to grade ≤1 or baseline due to agents administered, with exception of grade 2 fatigue, rash, and endocrinopathy successfully managed hormone replacement therapy, or alopecia or stable neuropathy, unless approved by the investigational new drug (IND) Sponsor.
* Patients with corrected QT interval (QTc) prolongation > 470 ms according to Fridericia formula.
* Patients receiving potent inducers of Cytochrome P450 3A (CYP 3A4/5) (including apalutamide, carbamazepine, enzalutamide, mitotane, phenytoin, rifampin and St. John's Wort) that cannot be discontinued at least 14 days prior to Cycle 1 Day 1.
* Known sensitivity to or history of allergic reactions attributed to compounds of similar chemical or biologic composition of DRP-104 or durvalumab.
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Has a pulse oximetry of <92% on room air or is on supplemental home oxygen.
* Active or untreated brain metastases or leptomeningeal metastases.
* Uncontrolled intercurrent active medical and/or psychiatric illness/social psychosocial problems that that would limit compliance with study requirements.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding.
* Has a known history of Human Immunodeficiency Virus (HIV)/AIDS.
* Has active hepatitis B. Patients with chronic or acute hepatitis B virus (HBV) infection .
* Have had evidence of active or acute diverticulitis, intra-abdominal abscess, or GI obstruction which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study.
* Patient is unwilling or unable to follow the study schedule for any reason.
* Patient is at the time of signing informed consent a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Evidence of clinical ascites.
* Participants a with history of prior unacceptable and/or life-threatening toxicities attributed to anti-programmed death-receptor 1 (PD1) or anti-PD-L1 (anti-programmed death-receptor 1) therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Prior allogeneic stem cell transplantation or organ transplantation.
* Has a diagnosis of immunodeficiency.
* Systemic corticosteroids at immunosuppressive doses.
* Patients who have had either of the following procedures or medications within 4 weeks prior to initiation of study treatment:
* Any live, attenuated vaccine
* Allergen hypo sensitization therapy in the last 2 weeks

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing drug-related adverse events (AEs) requiring treatment discontinuation | 4 years
  When calculating the incidence of AEs, each AE (as defined by NCI Common Terminology Criteria for Adverse Events [CTCAE] v5.0) will be counted only once for a given subject.
Objective response rate (ORR) using immune Response Evaluation Criteria for Solid Tumors (RECIST 1.1) | 4 years
  ORR is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) to DRP-104 (glutamine antagonist) in combination with duvalumab, based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30percent decrease in sum of diameters of target lesions, progressive disease (PD) is >20percent increase in sum of diameters of target lesions, stable disease (SD) is <30percent decrease or <20percent increase in sum of diameters of target lesions.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 4 years
  PFS is defined as the number of months from the date of first treatment to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Progression will be censored at the date of the last scan for subjects without documentation of disease progression at the time of analysis. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Overall survival (OS) | 4 years
  OS is defined as the number of months from the first dose of study treatment to death from any cause or end of follow-up. OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis. Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Baretti, MD, Principal Investigator — SKCCC • Johns Hopkins Medical Institution
Locations (1):
- Johns Hopkins SKCCC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No